CLINICAL TRIAL: NCT04293276
Title: Study to Evaluate the Efficacy and Safety of CDK4/6 Inhibitor SHR6390 Combined With Pyrotinib in the Treatment of HER2-positive Advanced Breast Cancer
Brief Title: Study to Evaluate the Efficacy and Safety of SHR6390 Combined With Pyrotinib in HER2+ Advanced Breast Cancer
Acronym: DAP-Her-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR BLTN 014
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Patients with HER2 positive breast cancer will receive Pyrotinib in combination with SHR6390(at protocol defined dose levels) orally until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Pyrotinib; Drug: SHR6390

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib Tablets
Drug: SHR6390 — SHR6390 Tablets

SUMMARY:
The main purpose of this study was to observe the efficacy and safety of treatment with pyrotinib and CDK4/6 inhibitor SHR6390 for HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Local recurrent or metastatic breast cancer suitable for chemotherapy, confirmed histologically.
* HER2-positive breast cancer(according to 2018 ASCO/CAP HER2 test guideline).
* Patients with HER2-positive metastatic breast cancer who had received ≤ 1-line treatment in the past;
* 18-70 years old;
* ECOG PS 0-1;
* Life expectancy is not less than 12 weeks;
* At least one measurable lesion according to RECIST 1.1;
* ANC ≥ 2.0×10^9/L, PLT ≥ 100×10^9/L, Hb ≥ 90 g/L; TBIL≤1.5ULN; ALT and AST≤3×ULN(ALT and AST≤5×ULN if liver metastasis); BUN and Cr≤1.5×ULN;
* LVEF ≥ 50% and QTc≤470 ms.

Exclusion Criteria:

* Patients with symptomatic brain metastasis;
* Unable to swallow, chronic diarrhea and intestinal obstruction, there are many factors affecting drug use and absorption;
* patient who received radiotherapy, chemotherapy, surgery (excluding local puncture) or molecular targeted therapy within 4 weeks before admission; those who received anti-tumor endocrine therapy after screening period;
* Participated in other drug clinical trials within 4 weeks before admission;
* Tyrosine kinase inhibitors targeting HER2 (Neratinib, Lapatinib, pyrotinib, etc.) have been used or are being used in the past;
* Other malignant tumors, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma, have been diagnosed in the past five years;
* A history of immunodeficiency, including HIV positive, HCV, or other acquired, congenital immunodeficiency disorders, or organ transplantation, is known;
* Has suffered from any heart disease;
* Female patients during pregnancy and lactation, fertile women with positive baseline pregnancy tests or women of childbearing age who are unwilling to take effective contraceptive measures throughout the trial;
* According to the judgement of the researchers, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of research (including, but not limited to, severe hypertension, severe diabetes, active infections, etc.);
* Moderate infection occurs within 4 weeks before the first administration (e.g. intravenous drip of antibiotics, antifungal or antiviral drugs according to clinical criteria), fever(> 38.5 ℃) of unknown origin occurs during the screening period/before the first administration;
* Researchers believe that patients are not suitable for any other situation in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
ORR | From the start of treatment to Disease Progress, assessed up to 2 years
  ORR by investigator using RECIST Guideline (Version 1.1)

SECONDARY OUTCOMES:
Adverse Events | from the first drug administration to 30 days from the last dose, assessed up to 2 years
  The number of patients experiencing any adverse events (AE) during the study time
PFS | up to 2 years
  Progression-Free Survival
OS | up to 2 years
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Professor, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Yan M, Niu L, Lv H, Zhang M, Wang J, Liu Z, Chen X, Lu Z, Zhang C, Zeng H, Zhao S, Feng Y, Sun H, Li H. Dalpiciclib and pyrotinib in women with HER2-positive advanced breast cancer: a single-arm phase II trial. Nat Commun. 2023 Oct 7;14(1):6272. doi: 10.1038/s41467-023-41955-7. PMID 37805496